CLINICAL TRIAL: NCT01662661
Title: A Phase I, Open-Label, Randomized, 2-way Crossover Study in Healthy Subjects to Assess the Relative Bioavailability of a Single Oral Dose of JNJ-47910382 Formulated as a Tablet and as a Suspension
Brief Title: A Study to Compare the Bioavailability of JNJ-47910382 Formulated as a Tablet and as Suspension in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR100881; 47910382HPC1004 (Other: Janssen R&D Ireland); 2012-002341-38 (EudraCT Number)
Record Dates: First submitted 2012-08-08; First posted 2012-08-10 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Healthy Participants
Keywords: Healthy participants; Hepatitis C; Relative bioavailability; Bioavailability; Pharmacokinetics; JNJ-47910382
MeSH Terms: conditions — Hepatitis C | interventions — Suspensions; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm AB (Experimental): Treatment A: 200 mg dose of JNJ-47910382 formulated as a suspension followed by Treatment B: 200 mg JNJ-47910382 formulated as an uncoated tablet, administered on Day 1.
  Interventions: Drug: JNJ-47910382 (suspension); Drug: JNJ-47910382 (tablet)
- Arm BA (Experimental): Treatment B: 200 mg JNJ-47910382 formulated as an uncoated tablet followed by Treatment A: 200 mg dose of JNJ-47910382 formulated as a suspension, administered on Day 1.
  Interventions: Drug: JNJ-47910382 (suspension); Drug: JNJ-47910382 (tablet)

INTERVENTIONS:
Drug: JNJ-47910382 (suspension) — Type=exact number, unit=mg, number=200, form=suspension, route=oral. JNJ-47910382 administered on Day 1.
Drug: JNJ-47910382 (tablet) — Type=exact number, unit=mg, number=200, form=tablet, route=oral. JNJ-47910382 administered on Day 1.

SUMMARY:
The purpose of this study is to assess the relative bioavailability (the degree to which the study medication becomes available in the blood circulation) of JNJ-47910382, given as an uncoated tablet and as a suspension, after a single oral dose of 200 mg in healthy adult participants under fed conditions.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), randomized (the study medication is assigned by chance), 2-way crossover study (method used to switch participants from one treatment arm to another in a clinical study) to compare the oral bioavailability of JNJ-47910382 formulated as an uncoated tablet and as a suspension, in healthy participants. The study consists of 3 phases, including, a screening phase, an open-label treatment phase, and a follow up phase. The screening phase will be within 21 days before administration of the first dose of study medication. After screening, participants will be randomized according to a classical 2 sequence (ie, treatment sequence AB [where the participants will first receive treatment A and then treatment B] and sequence BA [where the participants will first receive treatment B and then treatment A]), 2-period crossover design to receive the study medication in the treatment phase. In each session (Session 1 or Session 2), participants will receive either Treatment A: 200 mg dose of JNJ-47910382 formulated as a suspension, or Treatment B: 200 mg JNJ-47910382 formulated as an uncoated tablet. There will be a washout period (period when participant is not receiving any study medication) of at least 7 to 14 days between the 2 sessions. The follow up phase will include 2 follow up visits after intake of study medication in last treatment session. Safety evaluations for adverse events, clinical laboratory tests, electrocardiogram, vital signs, physical examination, and specific toxicities will be monitored throughout the study. The duration of the study will be at least 11 to 18 days (screening and follow up phase not included).

ELIGIBILITY:
Inclusion Criteria:

* Must be healthy on the basis of physical examination, medical history, vital signs and the results of blood biochemistry, hematology and coagulation tests and a urinalysis performed (at screening)
* Must have a triplicate 12-lead electrocardiogram consistent with normal cardiac conduction and function
* Must be a non-smoker for at least 3 months prior to selection
* If a female, must be postmenopausal or surgically sterile
* Female participants must have a negative serum pregnancy test (at screening)

Exclusion Criteria:

* Had a past history of heart arrhythmias, history of risk factors for Torsade de Pointes syndrome (an uncommon and distinctive form of polymorphic ventricular tachycardia characterized by a gradual change in the amplitude and twisting of the QRS complexes around the isoelectric line on the electrocardiogram) or having low potassium levels in the blood
* History or suspicion of alcohol, barbiturate, amphetamine, recreational or narcotic drug use that could impact compliance to protocol requirements and/or safety
* Hepatitis A, B or C infection (at screening)
* A positive human immunodeficiency virus type 1 or 2 (HIV-1 or HIV-2) test (at screening)
* Have a positive urine drug test or alcohol breath test (at screening)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2012-07; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | Day 1 (0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 12.0, 16.0 hours), Day 2 (24, 36 hours), Day 3 (48 hours), and Day 4 (72 hours)
Time to reach the maximum plasma concentration (Tmax) | Day 1 (0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 12.0, 16.0 hours), Day 2 (24, 36 hours), Day 3 (48 hours), and Day 4 (72 hours)
Area under the plasma concentration-time curve (AUC) | Day 1 (0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 12.0, 16.0 hours), Day 2 (24, 36 hours), Day 3 (48 hours), and Day 4 (72 hours)

SECONDARY OUTCOMES:
Number of participants with adverse events | Up to 58 days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Antwerp, Belgium